CLINICAL TRIAL: NCT02279290
Title: Using CBT to Probe Psychobiobehavioral Resilience to Post-trauma Psychopathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Alyson Zalta, Assistant Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K23MH103394 (NIH)
Record Dates: First submitted 2014-10-22; First posted 2014-10-31 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Anxiety; Depression
Keywords: Childhood trauma
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Mind Intervention (HMI) (Experimental): This intervention will focus on teaching individuals a way to manage acute and chronic stressors more effectively.
  Interventions: Behavioral: Healthy Mind Intervention (HMI)
- Healthy Body Intervention (HBI) (Active Comparator): This intervention will focus on important health-related topics.
  Interventions: Behavioral: Healthy Body Intervention (HBI)

INTERVENTIONS:
Behavioral: Healthy Mind Intervention (HMI) — Healthy Mind Intervention (HMI) is a flexible cognitive-behavioral resilience building program. Participants will receive 8 weekly, 60-minute individual sessions of HMI. In HMI, participants will be able to select 3 areas of resilience that they want to work on.
  Arms: Healthy Mind Intervention (HMI)
Behavioral: Healthy Body Intervention (HBI) — The 8 weekly, 60-minute individual sessions will include the following topics: the mind-body connection, nutrition, exercise, unhealthy substances, sleep, preventing illness, and preventive care. Each session is spent providing didactic information on these topics and strategies for how to engage in behavior change in these areas.
  Arms: Healthy Body Intervention (HBI)

SUMMARY:
This randomized controlled trial uses a modularized cognitive behavioral resilience training (MCBRT) intervention to probe risk and resilience mechanisms linked to post-trauma psychopathology. Ninety participants with a history of interpersonal trauma during childhood or adolescence and mild to moderate distress will be randomized to MCBRT or a health education control condition. The primary aims of this proposal are to examine whether individuals who receive MCBRT demonstrate increases in psychological resilience, biological resilience, and extinction learning compared to those in the control group. This study will also explore associations between these psychobiobehavioral risk and resilience factors.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. fluent in English
3. history of childhood interpersonal trauma (e.g., sexual assault, physical assault, witnessing assault before age 18)
4. mild to moderate distress indicated by a score of 10-20 on the depression scale, 8-14 on the anxiety scale, or 15-25 on the stress scale of the DASS-21.

Exclusion Criteria:

1. severe distress indicated by a score >20 on the depression scale, >14 on the anxiety scale, or >25 on the stress scale of the DASS-21
2. DSM-5 criterion A trauma in the past month
3. color blindness based on self-report (because of inability to complete the fear conditioning task)
4. auditory impairment based on audiometer screening (because of inability to complete the fear conditioning task)
5. lifetime psychotic or bipolar disorder
6. substance abuse or dependence within past 6 months
7. concurrent psychotherapy initiated within 3 months of randomization
8. ongoing psychotherapy of any duration directed toward treatment of trauma-related psychopathology (e.g., CBT)
9. must be on a stable dose of psychotropic or adrenergically-active medications (e.g., beta blockers) for at least 6 weeks prior to eligibility screening
10. mental retardation or significant cognitive impairment
11. serious medical illness or instability for which hospitalization may be likely within the next year
12. significant suicidal ideation indicated by "yes" on Columbia Suicide Severity Rating Scale item 4 (active suicidal ideation with some intent to act) or enacted suicidal behaviors within 6 months prior to eligibility
13. current legal actions related to trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Psychological resilience outcomes include emotion regulation (DERS), hardiness (CD-RISC), optimism (LOT-R), perceived control (SMS), social support (MSPSS), and task-oriented coping (CISS-SFT). | 0 - 9 weeks
  Difference between the interventions in the change of psychological resilience from pre to post intervention.
Biological resilience outcomes include neuropeptide Y [NPY], dehydroepiandrosterone [DHEA], allopregnanolone [ALLO] taken from a blood draw. | 0-9 weeks
  Difference between the interventions in the change of biological resilience from pre to post intervention.
Extinction learning will be analyzed using the fear potentiated startle data from a fear conditioning paradigm. | 0-9 weeks
  Difference between the interventions in the change of extinction learning from pre to post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Alyson K Zalta, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

DOCUMENTS (1):
  • Informed Consent Form (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT02279290/ICF_000.pdf